CLINICAL TRIAL: NCT00966563
Title: Mangafodipir as an Adjunct to Percutaneous Coronary Intervention in Acute Myocardial Infarction (MANAMI)
Brief Title: Mangafodipir as an Adjunct to Percutaneous Coronary Intervention
Acronym: MANAMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egetis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MANAMI PP01-09
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Myocardial Infarction
Keywords: Mangafodipir; Primary Percutaneous Coronary Intervention; Myocardial infarction; Troponin; CK-MB; Magnetic Resonance Imaging
MeSH Terms: conditions — Myocardial Infarction | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mangafodipir treatment (Active Comparator): Treatment will be undertaken with a ready-to use investigative drug formulation identical to what is in diagnostic use as a contrast medium for MRI. Formulation content: MnDPDP 10 mmol/ml.
  Interventions: Drug: Mangafodipir
- NaCl 0.9% (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mangafodipir — Administered dose: 2 µmol/kg b.w. Administration form: Ready-to-use formulation (solution). Mangafodipir or placebo (0.2 ml/kg b.w.) will be administered as an intravenous (iv.) infusion over 2-5 min prior to reopening of occluded coronary artery during PCI
  Other Names: Teslascan
  Arms: Mangafodipir treatment
Drug: Placebo
  Arms: NaCl 0.9%

SUMMARY:
The present feasibility study is designed to find out whether pre-treatment with the compound mangafodipir (PP-099) provides an additional reduction in myocardial infarct size in patients treated with primary percutaneous coronary intervention (PCI) during acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
Mangafodipir, manganese (Mn) dipyridoxyl diphosphate (MnDPDP) and its lipophile metabolite Mn dipyridoxyl diethylene diamide (MnPLED), are catalytic antioxidants and iron chelators. In preclinical studies these agents reduce oxidative stress induced injuries related to chemotherapy of cancer and to reperfusion/reoxygenation of ischemic/hypoxic myocardium. Accordingly, in an in vivo pig model of AMI metabolite MnPLED applied at end of ischemia and during reperfusion reduced myocardial infarct size by 55 %. Mangafodipir most likely activates salvage pathways and prevents lethal reperfusion injuries.

Other advantages are that mangafodipir is already approved as a contrast agent for MRI of liver, and that the experience for more than a decade reveals a high safety with minor and tolerable side-effects.

The present study will include 20 patients treated for their first documented AMI. They will after admission to hospital undergo primary PCI. Reopening of an occluded coronary artery will be preceded by iv. infusion of mangafodipir or placebo in two groups , each consisting of 10 patients. The primary endpoint will be release to plasma of commonly accepted biomarkers of myocardial injury (Troponin T and CK-MB) measured at admission and 6 hours after PCI. The secondary endpoints include the accumulated release of plasma biomarkers over 48 hours and direct measurement of the final myocardial infarct size at 6-10 weeks after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Males 40-80 and females 50-80 years with first severe coronary attack
2. Chest pain up to 6 hours.
3. T segment elevation (≥ 0.2 mV in two neighbouring anterior and inferior wall leads.
4. Decided for treatment by primary PCI.
5. TIMI grade 0 flow in the occluded LAD or RCA artery
6. Written informed consent.

Exclusion Criteria:

1. Previous coronary artery bypass operation.
2. Previous AMI.
3. Chest pain more than 6 hours.
4. Angina within 48 hours before admission.
5. Cardiac arrest and cardiogenic shock.
6. Occlusion of the left main stem, circumflex and right coronary arteries at angiography.
7. Known hypersensitivity to mangafodipir (as contrast agent for MRI).
8. Received mangafodipir ≤ 5 weeks before admission
9. History of prior serious allergic or pseudo-allergic reaction
10. Severely reduced liver or renal function
11. Any other serious illness or medical condition
12. Fertile females
13. Phaeochromocytoma

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction of myocardial infarct size assessed by biomarker release to plasma | Before and at 2 days after PCI

SECONDARY OUTCOMES:
Reduction of myocardial infarct size assessed by biomarker release to plasma and by magnetic resonance imaging (MRI) of the heart. | Accumulated biomarker release over 48 hours after PCI; MRI at 6-10 weeks after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Erik Karlsson, MD, PhD, Principal Investigator — Department of Internal Medicine, County Hospital Ryhov, SE-551 85 Jönköping, Sweden
Locations (1):
- Department of Internal Medicine, County Hospital Ryhov, Jönköping, Sweden

REFERENCES:
- [Background] 1. Piot C, Croisille P, Staat P, Thibault H, Rioufol G et al. Effect of cyclosporine on reperfusion injury in acute myocardial infarction. New Engl J Med 2008; 359: 473-481. 2. Yellon DM, Hausenloy DJ. Mechanisms of disease: Myocardial reperfusion injury. New Engl J Med 2007; 357: 1121-1135. 3. Karlsson JOG, Brurok H, Eriksen M, Towart R, Toft KG, Moen O, Engebretsen B, Jynge P and Refsum H. Cardioprotective effects of the MR contrast agent MnDPDP and its metabolite MnPLED upon reperfusion of the ischemic porcine myocardium. Acta Radiologica 2001;42:540-547. 4. Brurok H, Ardenkjær-Larsen JH, Hansson G, Skarra S, Berg K, Karlsson JOG, Jynge P. Manganese dipyridoxyl diphosphate: MRI contrast agent with antioxidative and cardioprotective properties. Biochem Biophys Res Commun 1999;254:768-772. 5. Karlsson JOG, Brurok H, Towart R, Jynge P. Letter to the Editor. The magnetic resonance imaging contrast agent mangafodipir exerts antitumor activity via a previously described superoxide mimetic activity. Cancer Res 2006;66:598. 6. MANFOL. Mangafodipir as an adjunct to FOLFOX6 chemotherapy in colon cancer stage Duke's C. Study NCT00671996. 2008. 7. Skjold A, Amundsen BH, Wiseth R, Støylen A, Haraldseth O, Larsson HB, Jynge P. Manganese dipyridoxyl-diphosphate (MnDPDP) as a viability marker in patients with myocardial infarction. J Magn Reson Imaging 2007; 26: 720-727. 8. Jynge P, Brurok H, Asplund A, Towart R, Refsum H, Karlsson JOG. Cardiovascular safety of MnDPDP and MnCl2. Acta Radiol 1997;38:740-749. 9. Karlsson JOG, Mortensen E, Pedersen HK, Sager G, Refsum H. Cardiovasular effects of MnDPDP and MnCl2 in dogs with acute ischemic heart failure. Acta Radiol 1997;38:750-758.